CLINICAL TRIAL: NCT00817557
Title: Use of Loteprednol for Contact Lens Intolerance and Dryness
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hom, Milton M., OD, FAAO (Individual)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Milton M. Hom, OD, FAAO., Private Practice
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 05
Record Dates: First submitted 2009-01-02; First posted 2009-01-06 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Contact Lenses Dryness
Keywords: Contact lenses; Loteprednol; Effect on CL dryness
MeSH Terms: interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Loteprednol (Active Comparator): Loteprednol BID
  Interventions: Drug: Loteprednol
- Rewetter (Placebo Comparator): Rewetter BID
  Interventions: Other: Rewetter

INTERVENTIONS:
Drug: Loteprednol — Anti-inflammatory
  Arms: Loteprednol
Other: Rewetter
  Arms: Rewetter

SUMMARY:
Study of the effects of Loteprednol on CL dryness

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and over inclusive.
2. Males or females
3. Any race or ethnic background
4. CL history- experienced intolerance and either switched solutions or lenses without satisfactory relief.
5. Patient is in generally good & stable overall health.
6. Patient likely to comply with study guidelines & study visits.
7. Informed consent signed.
8. OSDI score 18 or higher while wearing lenses
9. Unsatisfactory wearing time with contact lenses

Exclusion Criteria:

1. Corneal refractive surgery within 6 months of this study.
2. Contact lens use on day of examination.
3. Corneal ectasia.
4. Current use of Restasis
5. Intra-ocular surgery within 6 months or ocular laser surgery within 6 months.
6. Pregnant or lactating women.
7. Ocular pathology (includes glaucoma and cataract) which could impact results and/or place patient at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Wearing time | 28 days

SECONDARY OUTCOMES:
OSDI | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Milton M Hom, OD FAAO, Principal Investigator — Private Practice
Locations (1):
- Milton M. Hom, OD, FAAO., Azusa, California, United States